CLINICAL TRIAL: NCT05831969
Title: Lenalidomide to Reverse Drug Resistance After Lenvatinib Combined With PD-1 Inhibitors in the First-line Treatment of Advanced HCC ：a Prospective, Exploratory, Single-arm, Open-label, Multi-center Clinical Study
Brief Title: Lenalidomide to Reverse Drug Resistance After First-line Treatment of Advanced HCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenyang Tenth People's Hospital (Other)
Collaborators: Beijing Tsinghua Changgeng Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dream-004
Record Dates: First submitted 2023-04-16; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-03

CONDITIONS: Advanced HCC
Keywords: lenalidomide; Drug resistance
MeSH Terms: interventions — Lenalidomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lenalidomide (Experimental): lenalidomide be used after Lenvatinib combined with PD-1 inhibitors in the first-line treatment
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide: 10mg/d, 1-21d/28d orally; until disease progression or intolerable adverse reactions.

SUMMARY:
The ORR of the lenvatinib combination (lenvatinib combined with PD-1 inhibitor) was largely similar to that of the "A+T" combination (bevacizumab and atelelizumab). The disease control rate (DCR) for the combination of lenvatinib was 88%, demonstrating the efficacy of lenvatinib in combination with immunotherapy. However, progression to second-line therapy after first-line treatment for advanced HCC still faces many challenges.

In our clinical practice and review of the literature, we focused on lenalidomide showing some efficacy in second-line treatment of advanced HCC. Lenalidomide is a new generation derivative of thalidomide, which has dual anti-angiogenic and immunomodulatory anti-tumor effects. Lenalidomide may have the potential to reverse drug resistance and increase the efficacy of synergistic immune-targeted therapy. Based on the preliminary data of its effectiveness in the second-line treatment of advanced HCC alone or in combination with TKI, we propose to conduct a prospective, exploratory, single-arm, open, multicenter phase II clinical study of advanced HCC PD-1 inhibitor in combination with lenvatinib after progression of first-line treatment, to initially evaluate the efficacy and safety of this regimen.

DETAILED DESCRIPTION:
Advanced primary hepatocellular carcinoma (HCC) has entered a new phase of clinical research and patient outcomes with the continued availability of new targeted agents and immune checkpoint inhibitors. More notable are lenvatinib in combination with PD-1 inhibitor regimens and the data that continue to emerge from these studies.

The 2020 ASCO GI published the Study117, a phase Ib clinical study of lenvatinib in combination with Nivolumab for the first-line treatment of unresectable hepatocytes. The study was an open phase Ib study that enrolled 30 patients, 17 with BCLC- stage B and 13 with BCLC- stage C. In the ITT population, the median age of patients was 70 years (range: 36-81 years) and 24 (80%) were male. 28 patients with ECOG performance status of ECOG 0 and 1 patient with ECOG 2 were enrolled. Enrolled patients received lenvatinib 12 mg (weight ≥60 kg) or 8 mg (weight <60 kg) orally once daily and in combination with Nivolumab 240 mg intravenously once every 2 weeks. The study results were impressive, with an investigator-assessed overall complete remission rate of 10% CR, a partial remission rate of 66.7% PR, an objective remission rate of 76.7% ORR, and a disease control rate of 96.7% DCR.

The ORR of the lenvatinib combination (lenvatinib in combination with PD-1 inhibitor) was generally similar to that of the "A+T" combination (bevacizumab and atelelizumab). The disease control rate (DCR) for the lenvatinib combination was 88%, indicating the efficacy of lenvatinib in combination with immunotherapy.

However, there are still many challenges in progressing to second-line therapy after first-line treatment for advanced HCC. The first is the limited efficacy of second-line treatment options recommended by NCCN guidelines.

The RESORCE study showed that single-agent regorafenib after sorafenib failure treated patients with Child-Pugh class A liver function had a higher mOS (10.6 months vs. 7.8 months) and mPFS (3.1 months vs. 1.5 months) than the placebo group. the CELESTIAL study showed that single-agent cabozantinib for patients previously treated with sorafenib in patients with HCC who were eligible for progression after at least first-line systemic therapy, 707 patients were randomly assigned in a 2:1 ratio to receive either cabozantinib (60 mg, QD) or placebo. OS was significantly longer in the cabozantinib group (10.2 months vs. 8.0 months, P=0.005). mPFS was 5.2 months vs. 1.9 months, respectively (P<0.001); ORR was 4% and <1%, respectively (P=0.009). A randomized, double-blind, placebo-controlled, global phase III clinical study of advanced HCC patients with elevated AFP after first-line failure of sorafenib enrolled 292 HCC patients with failed sorafenib and baseline AFP ≥ 400ng/ml who were randomized to receive either Ramucirumab (8mg/kg) or placebo in a 2:1 ratio. Compared with placebo, ramolutumab improved patients' mOS (8.5 months vs. 7.3 months, P=0.019 9) and mPFS (2.8 months vs. 1.6 months, P<0.0001) and reduced the risk of death by 29%; while ORR was 4.6% and 1.1%, respectively (P=0.115 6).The CheckMate-040 study [ 7] opened a phase II study of a dual immune combination therapy strategy with Nivolumab in combination with Ipilimumab) for the second-line treatment of advanced HCC, enrolling patients with advanced HCC intolerant or progressing on sorafenib therapy, with 33% (16/49; 95% CI 20 to 48) responding to immune combination therapy; BICR was assessed according to RECIST v1.1 criteria, with 8% (4 /49) achieved CR and 24% (12/49) PR; DOR ranged from 4.6 months to 30.5 months, of which 88% lasted at least 6 months, 56% at least 12 months, and 31% at least 24 months. However, all of the above studies were done after failure of sorafenib alone, and there are no effective treatment options for progression beyond targeted combination immunotherapy.

Due to the higher ORR of lenvatinib in combination with PD-1 antibody and the absence of risk of lethal bleeding, lenvatinib in combination with PD-1 antibody for advanced hepatocellular carcinoma is used by most physicians in real-world applications in China with good results, but there is no effective second-line treatment option for patients who fail lenvatinib in combination with PD-1 antibody, so our study explores whether lenalidomide can reverse lenvatinib patients who are resistant to lenvatinib in combination with PD-1 antibodies.

The phase II clinical study by the Brown University Oncology Group showed that lenalidomide was used as second-line treatment for advanced hepatocellular carcinoma, with 6 of 40 patients (15%) having a partial response and 2 patients (5%) having progression-free survival of 36 and 32 months, respectively, with a median progression-free survival of 3.6 months and a median overall survival of 7.6 months. Lenalidomide is safe and effective in the treatment of patients with Child-Pugh A and B cirrhosis [8]. A study in Taiwan found lenalidomide to be active in patients with advanced HCC with a good safety profile. The remission rate of advanced HCC progressing on lenalidomide monotherapy with sorafenib was 13% and the disease control rate was 53%. the 6-month progression-free survival rate was 9.1%. Median progression-free survival and overall survival were 1.8 months and 8.9 months, respectively. Early AFP response was significantly associated with higher disease control (76% vs 22%, P=0.001) and longer progression-free survival (P=0.020) . A study showed that apatinib combined with lenalidomide for advanced primary hepatocellular carcinoma improved treatment outcome and quality of life, with an overall effective rate of 89.7% vs 79.6% in the apatinib combined with lenalidomide treatment group compared to the apatinib alone group, respectively (P<0.01), while reducing the incidence of proteinuria, hypertension, hand-foot syndrome, diarrhea, and malaise.

Lenalidomide, a new generation derivative of thalidomide, has dual anti-angiogenic and immunomodulatory antitumor effects . Lenalidomide binds to its substrate CRBN and forms a copolymer with ubiquitinase E3, which degrades lymphocyte development-related tumor factors IKZF 1 and IKZF 3 through ubiquitination. degradation of IKZF 1 inhibits the binding of downstream substrate IRF4 to Myc and its expression, thus achieving antitumor effects; degradation of IKZF3 factor promotes the proliferation of effector T cells and NK cells and induces the secretion of anti-tumor factors such as IFNγ by effector T cells and NK cells. The degradation of IKZF3 factor can promote the proliferation of effector T cells and NK cells, and can induce the secretion of anti-tumor factors such as IFNγ by effector T cells and NK cells.

Recent studies have confirmed that lenalidomide can reverse PD-1 inhibitor resistance, and a study from the group of Cang Yong at the University of Science and Technology Shanghai found that PD-1 inhibitors require CD28 co-stimulatory receptors to promote CD8+ T cell activity and cytotoxicity. However, during depleted T cells and immune senescence, CD28 expression is frequently inactivated leading to PD-1 inhibitor resistance, which limits the antitumor efficacy of PD-1 immunotherapy. This study shows that lenalidomide restores the antitumor activity of cd28 -deficient CD8+ T cells after PD-1 resistance. Lenalidomide can target CRBN ubiquitin ligase to degrade Ikzf1 and Ikzf3 in T cells and release paracrine interleukin-2 (IL-2) and intracellular Notch signaling that are required to activate CD8+ T cells in tumors and inhibit tumor growth via PD-1 blockade. The findings suggest that PD-1 immunotherapy of solid tumors in a CD28- T cell infiltration-rich state could benefit from a combination of lenalidomide reversal of drug resistance.

In view of the above, we believe that lenalidomide may have the potential to reverse drug resistance and increase efficacy with synergistic immune-targeted therapy. Based on its preliminary efficacy data in second-line treatment of advanced HCC alone or in combination with TKI, we propose to conduct a prospective, exploratory, single-arm, open, multicenter phase II clinical study of advanced HCC PD-1 inhibitor in combination with lenvatinib after progression to first-line therapy plus lenalidomide to preliminarily evaluate the efficacy and safety of this regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to sign a written informed consent;
2. Age ≥ 18 and ≤ 75 years old on the day of signing the informed consent form;
3. Locally advanced hepatocellular carcinoma, clinical diagnosis of hepatocellular carcinoma by histology/cytology, imaging (enhanced MRI or enhanced CT or PET-CT);
4. Advanced metastatic and/or unresectable HCC progresses after combination therapy with lenvatinib combined with PD-1 inhibitors (must be domestically approved for use in liver cancer);
5. Eastern Cooperative Oncology Group (ECOG) physical status score is 0 or 1;
6. Liver function in line with Child-Pugh A grade (score 5-6 points);
7. Hepatitis B surface antigen detection is required before enrollment. For patients who are confirmed to have hepatitis B, antiviral drugs should be started 1 week before treatment;
8. During the study screening period, patients must be tested for hepatitis C virus (HCV) RNA status. This study allowed for the study of patients with untreated chronic HCV infection. In addition, patients who have been cured of hepatitis C can be included in this study, but the hepatitis C treatment should be completed for more than 4 weeks at the time of enrollment;
9. The main organ functions are basically normal and meet the following requirements:

   Bone marrow: absolute neutrophil count ≥1.5×109/L, platelet ≥50×109/L, hemoglobin ≥90g/L.

   Liver: total bilirubin ≤ 2 times the upper limit of normal (ULN), aspartate aminotransferase and alanine aminotransferase ≤ 5 × ULN, albumin ≥ 29 g/L.

   Kidney: serum creatinine ≤1.5×ULN, or creatinine clearance ≥50mL/min. Coagulation function: international normalized ratio (INR) ≤ 2, and activated partial thromboplastin time (APTT) ≤ 1.5 times ULN.
10. The expected survival time is more than 3 months;
11. Patients with other malignant tumors have lived disease-free for more than 2 years after initial treatment (such as non-melanoma skin cancer or cervical cancer in situ);
12. Women of childbearing age must agree to use effective contraception for at least 4 weeks before enrollment in the study, during the study and within 4 weeks after the withdrawal of the study drug. Women of childbearing potential require a serum pregnancy test within 72 hours of starting treatment. Male subjects must also use effective contraception during treatment and within 4 weeks of drug withdrawal. The spouse of the subject also needs to do a good job of contraception during the subject's participation in the study;
13. Did not participate in other clinical trials within 4 weeks before screening; those who failed to screen in other trials but met the requirements of this trial can be enrolled.

Exclusion Criteria:

1. Hypersensitivity to iridamine drugs;
2. Fibrolamellar or sarcomatoid HCC;
3. Mixed HCC-ICC;
4. Currently participating in and receiving other experimental treatments, or participating in a study of immune checkpoint inhibitors and receiving study treatment;
5. Previous solid organ transplantation, diagnosed as immunodeficiency, or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days before the first trial treatment;
6. Esophageal or gastric variceal bleeding within 3 months before enrollment;
7. Hepatic encephalopathy in the past 6 months, or obvious ascites at the time of enrollment;
8. Have a known history of active tuberculosis;
9. Hypersensitivity to PD-1 inhibitors;
10. The subject has other known aggressive malignant tumors at the same time (except for those who have no evidence of tumor recurrence after treatment and the duration is more than 2 years). Exceptions include: basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, low-risk prostate cancer, or cervical cancer in situ;
11. Patients with previous active autoimmune diseases requiring systemic treatment;
12. History or any evidence of known active non-infectious pneumonia;
13. Active infection requires systemic treatment;
14. People with known mental illness or substance abuse disorder;
15. Pregnant or lactating women;
16. Known human immunodeficiency virus (HIV) medical history (HIV 1/2 antibody);
17. Have been vaccinated with live vaccines within 30 days before starting the study treatment;
18. Those who suffer from high blood pressure and cannot be well controlled by antihypertensive drug treatment (systolic blood pressure>140mmHg, diastolic blood pressure>100mmHg); suffer from myocardial ischemia or myocardial infarction above CTCAE grade II, poorly controlled arrhythmia, And/or New York Heart Association (NYHA) class III~IV cardiac insufficiency;
19. Other conditions that the investigator believes prevent patients from participating in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2023-06-05 (Estimated); Primary Completion 2025-06-05 (Estimated); Study Completion 2025-10-05 (Estimated)

PRIMARY OUTCOMES:
ORR | up to approximately 24 months
  Defines the proportion of patients whose tumor volume shrinks to a prespecified value and is maintained for a minimum period of time. The RECIST 1.1 standard was adopted, including complete remission of CR and partial remission of PR.

SECONDARY OUTCOMES:
PFS | Randomization to the first occurrence of disease progression or death from any cause up to the clinical cut off date of June 5,2024
  PFS was defined as the time from randomization to the first occurrence of progressive disease (PD) or death from any cause whichever occurs first as determined by an IRF according to RECIST v1.1. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters on study (including baseline).
  In addition to the relative increase of 20%, the sum of diameters must also demonstrate an absolute increase of >/= 5 millimeters (mm).
OS | up to approximately 24 months
  Time from enrollment to death (for any reason);
DOR | up to approximately 18 months
  Time from the first CR or PR to disease progression after enrollment
Percentage of Participants With Adverse Events | Up to end of study (up to approximately 24 months
  An adverse event is any untoward medical occurrence in a subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jianhui Jia, M.B, Principal Investigator — Shenyang Tenth People's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Finn RS, Ikeda M, Zhu AX, Sung MW, Baron AD, Kudo M, Okusaka T, Kobayashi M, Kumada H, Kaneko S, Pracht M, Mamontov K, Meyer T, Kubota T, Dutcus CE, Saito K, Siegel AB, Dubrovsky L, Mody K, Llovet JM. Phase Ib Study of Lenvatinib Plus Pembrolizumab in Patients With Unresectable Hepatocellular Carcinoma. J Clin Oncol. 2020 Sep 10;38(26):2960-2970. doi: 10.1200/JCO.20.00808. Epub 2020 Jul 27. PMID 32716739
- [Background] IMbrave150: Exploratory Efficacy and Safety Results in Patients With Hepatocellular Carcinoma Without Macrovascular Invasion or Extrahepatic Spread Treated With Atezolizumab + Bevacizumab or Sorafenib. Gastroenterol Hepatol (N Y). 2021 Nov;17(11 Suppl 6):14-15. No abstract available. PMID 35611267
- [Background] Bruix J, Qin S, Merle P, Granito A, Huang YH, Bodoky G, Pracht M, Yokosuka O, Rosmorduc O, Breder V, Gerolami R, Masi G, Ross PJ, Song T, Bronowicki JP, Ollivier-Hourmand I, Kudo M, Cheng AL, Llovet JM, Finn RS, LeBerre MA, Baumhauer A, Meinhardt G, Han G; RESORCE Investigators. Regorafenib for patients with hepatocellular carcinoma who progressed on sorafenib treatment (RESORCE): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2017 Jan 7;389(10064):56-66. doi: 10.1016/S0140-6736(16)32453-9. Epub 2016 Dec 6. PMID 27932229
- [Background] Abou-Alfa GK, Meyer T, Cheng AL, El-Khoueiry AB, Rimassa L, Ryoo BY, Cicin I, Merle P, Chen Y, Park JW, Blanc JF, Bolondi L, Klumpen HJ, Chan SL, Zagonel V, Pressiani T, Ryu MH, Venook AP, Hessel C, Borgman-Hagey AE, Schwab G, Kelley RK. Cabozantinib in Patients with Advanced and Progressing Hepatocellular Carcinoma. N Engl J Med. 2018 Jul 5;379(1):54-63. doi: 10.1056/NEJMoa1717002. PMID 29972759
- [Background] Zhu AX, Kang YK, Yen CJ, Finn RS, Galle PR, Llovet JM, Assenat E, Brandi G, Pracht M, Lim HY, Rau KM, Motomura K, Ohno I, Merle P, Daniele B, Shin DB, Gerken G, Borg C, Hiriart JB, Okusaka T, Morimoto M, Hsu Y, Abada PB, Kudo M; REACH-2 study investigators. Ramucirumab after sorafenib in patients with advanced hepatocellular carcinoma and increased alpha-fetoprotein concentrations (REACH-2): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2019 Feb;20(2):282-296. doi: 10.1016/S1470-2045(18)30937-9. Epub 2019 Jan 18. PMID 30665869
- [Background] Yau T, Kang YK, Kim TY, El-Khoueiry AB, Santoro A, Sangro B, Melero I, Kudo M, Hou MM, Matilla A, Tovoli F, Knox JJ, Ruth He A, El-Rayes BF, Acosta-Rivera M, Lim HY, Neely J, Shen Y, Wisniewski T, Anderson J, Hsu C. Efficacy and Safety of Nivolumab Plus Ipilimumab in Patients With Advanced Hepatocellular Carcinoma Previously Treated With Sorafenib: The CheckMate 040 Randomized Clinical Trial. JAMA Oncol. 2020 Nov 1;6(11):e204564. doi: 10.1001/jamaoncol.2020.4564. Epub 2020 Nov 12. PMID 33001135
- [Background] Safran H, Charpentier KP, Kaubisch A, Mantripragada K, Dubel G, Perez K, Faricy-Anderson K, Miner T, Eng Y, Victor J, Plette A, Espat J, Bakalarski P, Wingate P, Berz D, Luppe D, Martel D, Rosati K, Aparo S. Lenalidomide for second-line treatment of advanced hepatocellular cancer: a Brown University oncology group phase II study. Am J Clin Oncol. 2015 Feb;38(1):1-4. doi: 10.1097/COC.0b013e3182868c66. PMID 23648434
- [Background] Shao YY, Chen BB, Ou DL, Lin ZZ, Hsu CH, Wang MJ, Cheng AL, Hsu C. Lenalidomide as second-line therapy for advanced hepatocellular carcinoma: exploration of biomarkers for treatment efficacy. Aliment Pharmacol Ther. 2017 Oct;46(8):722-730. doi: 10.1111/apt.14270. Epub 2017 Aug 17. PMID 28815645
- [Background] Richardson P, Anderson K. Immunomodulatory analogs of thalidomide: an emerging new therapy in myeloma. J Clin Oncol. 2004 Aug 15;22(16):3212-4. doi: 10.1200/JCO.2004.05.984. Epub 2004 Jul 12. No abstract available. PMID 15249587
- [Background] Lindner S, Kronke J. The molecular mechanism of thalidomide analogs in hematologic malignancies. J Mol Med (Berl). 2016 Dec;94(12):1327-1334. doi: 10.1007/s00109-016-1450-z. Epub 2016 Aug 5. PMID 27492707
- [Background] Guirguis AA, Ebert BL. Lenalidomide: deciphering mechanisms of action in myeloma, myelodysplastic syndrome and beyond. Curr Opin Cell Biol. 2015 Dec;37:61-7. doi: 10.1016/j.ceb.2015.10.004. Epub 2015 Nov 11. PMID 26512454
- [Background] Nicholas NS, Apollonio B, Ramsay AG. Tumor microenvironment (TME)-driven immune suppression in B cell malignancy. Biochim Biophys Acta. 2016 Mar;1863(3):471-482. doi: 10.1016/j.bbamcr.2015.11.003. Epub 2015 Nov 7. PMID 26554850
- [Background] Chong EA, Ahmadi T, Aqui NA, Svoboda J, Nasta SD, Mato AR, Walsh KM, Schuster SJ. Combination of Lenalidomide and Rituximab Overcomes Rituximab Resistance in Patients with Indolent B-cell and Mantle Cell Lymphomas. Clin Cancer Res. 2015 Apr 15;21(8):1835-42. doi: 10.1158/1078-0432.CCR-14-2221. Epub 2015 Jan 28. PMID 25632047
- See also: Related Info — http://pubmed.aaaib.top/32716739/
- See also: Related Info — http://pubmed.aaaib.top/35611267/
- See also: Related Info — http://pubmed.aaaib.top/27932229/
- See also: Related Info — http://pubmed.aaaib.top/29972759/
- See also: Related Info — http://pubmed.aaaib.top/30665869/
- See also: Related Info — http://pubmed.aaaib.top/33001135/
- See also: Related Info — http://pubmed.aaaib.top/23648434/
- See also: Related Info — http://pubmed.aaaib.top/28815645/
- See also: Related Info — http://pubmed.aaaib.top/15249587/
- See also: Related Info — http://pubmed.aaaib.top/27492707/
- See also: Related Info — http://pubmed.aaaib.top/26512454/
- See also: Related Info — http://pubmed.aaaib.top/26554850/
- See also: Related Info — http://pubmed.aaaib.top/25632047/
- See also: Related Info — https://med.wanfangdata.com.cn/Paper/Detail?id=PeriodicalPaper_gdyxyxb202003020&dbid=WF_QK
- See also: Related Info — https://med.wanfangdata.com.cn/Paper/Search?q=%E6%9D%A5%E9%82%A3%E5%BA%A6%E8%83%BA%E9%80%9A%E8%BF%87%E6%8A%91%E5%88%B6VEGF%E8%9B%8B%E7%99%BD%E8%A1%A8%E8%BE%BE%E6%8A%91%E5%88%B6%E4%BA%BA%E8%82%9D%E7%99%8C%E7%BB%86%E8%83%9ELM3%E7%9A%84%E8%BF%81%E7%A7%BB%E5%92%8C%E4%BE%B5%E8%A2%AD